CLINICAL TRIAL: NCT02446288
Title: A Pilot Study of the TMJ NextGeneration Compared to the DSG Relaxer for Reduction in Nocturnal Bruxism Episodes in Subjects Diagnosed With Sleep Bruxism
Brief Title: TMJ NextGen Pilot Study to Treat Subjects With Bruxism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cardiox Corporation (Industry)
Collaborators: TMJ Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMJ-1003
Record Dates: First submitted 2015-05-12; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMJ Next Generation (Active Comparator): The TMJ NextGeneration device consists of a pair of small, hollow ear inserts. These ear inserts are custom-fit to each subject's ear canals. They are constructed from methacrylate polymers - the same material as has been used in hearing aids. The devices rest in the outer third of the ear canal and have a small retraction post that allows for removal of the device from the ear. The devices conform to the shape of the individuals' ear canals when the jaw is in the open position and permit full passage of sound into each ear. The proposed mechanisms of action of the inserts are to support the TMJ and associated secondary musculature to reduce strain in the TMJ area and to provide cognitive awareness to the wearer regarding para-functional habits, i.e., jaw clenching.
  Interventions: Device: TMJ Next Generation
- DSG Relaxer (Active Comparator): The occlusal splint to be used in this study will be the DSG Relaxer™. The DSG Relaxer™ is a device that has been FDA cleared for the treatment of medically diagnosed migraine pain as well as migraine associated tension-type headaches and relieving bruxism and TMJ syndrome through the reduction of trigeminally innervated muscular therapy.
  Interventions: Device: DSG Relaxer

INTERVENTIONS:
Device: TMJ Next Generation
  Arms: TMJ Next Generation
Device: DSG Relaxer
  Arms: DSG Relaxer

SUMMARY:
The study is an open-label, prospective, multicenter, randomized, two treatment parallel, comparison study of the TMJ NextGeneration and DSG Relaxer in the reduction of nocturnal bruxism episodes in subjects diagnosed with sleep bruxism.

DETAILED DESCRIPTION:
The study will be conducted at multiple study centers in the U.S. Subjects will be enrolled in the trial for a period of 44 days. The study will consist of a screening period lasting up to 30 days, a device fitting period of 14 days, and a treatment period lasting 30 days. Subjects will visit the clinic three times during the screening period, followed by visits at Day 1, Day 14, and Day 44 of the study. Subjects will visit the sleep center once during the screening period (Day -1) and once during the treatment period (Day 43).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects at least 18 years of age;
2. Subject has had a diagnosis of sleep bruxism confirmed within the past 30 days;
3. Subject has an average of ≥ 1.25 bruxism episodes per hour of sleep based on two nights of screening Bruxoff™ evaluations;
4. Subject is able to read and understand the ICF and has voluntarily provided written informed consent;
5. Subject has a minimum of 26 remaining teeth;
6. Subject has an average of ≥ 1.25 bruxism episodes per hour of sleep based on the single-night screening sleep PSG evaluations.

Exclusion Criteria:

1. Subjects with any physical or behavioral disorder, which, in the opinion of the Principal Investigator, may interfere with the use of the device or compliance with the study protocol;
2. Subject has a significant respiratory disease that actively requires treatment;
3. Subject is taking antidepressant medication;
4. Subject has a significant sleep disorder that actively requires treatment, in addition to bruxism;
5. Subject is undergoing treatment for sleep apnea;
6. Subjects diagnosed with rheumatoid arthritis, osteoarthritis, osteoarthrosis, or another connective tissue disorder of the head/neck region;
7. Subjects who have had direct trauma to the jaw;
8. Subjects who have used an occlusal appliance to treat a TMD within the previous six months;
9. Subjects who have had prior TMJ or ear surgery;
10. Subjects who have a narrow ear canal or impression of the ear canal, which is prolapsed due to an anatomical shift or failure of the ear canal wall structure, or a canal that does not allow for the ear canal second turn to be identified;
11. Subjects with visible or congenital ear deformity as observed on targeted physical exam that does not allow for fitting of the study device;
12. Subjects who have taken a narcotic pain medication in the last seven days prior to Day 1 of the study;
13. Subjects who have a history of chronic ear pain unrelated to TMJ;
14. Subjects who have a history of ear drainage in the past six months;
15. Subjects who have active ear drainage, swelling, or redness as observed on targeted physical exam;
16. Subjects whom the investigator believes may not be an appropriate candidate for an intra-oral splint due to missing or poor quality dentition or untreated pain of dental origin (pulpal pain, pericoronitis of wisdom teeth, or similar conditions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the effectiveness of the TMJ NextGeneration to reduce nocturnal bruxism episodes in subjects experiencing sleep bruxism as determined by polysomnography. | 30 days

SECONDARY OUTCOMES:
The secondary objective of this study is to further establish the safety of the TMJ NextGeneration device as determined by adverse events. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Simon Blackburn, CCRA, Study Director — Cardiox Corporation